CLINICAL TRIAL: NCT06520943
Title: Comparison of Minimum Flow Desflurane Anesthesia With Respiratory Parameters and Blood Gas Analyses and Low Flow Desflurane Anesthesia in Robotic Assisted Laparoscopic Abdominal Surgery
Brief Title: Comparison of Minimum Flow and Low Flow Desflurane Anesthesia in Robotic Assisted Laparoscopic Abdominal Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Betül Güven, assoc. prof, Ankara City Hospital Bilkent
Other Study IDs: TABED1-24-72
Record Dates: First submitted 2024-07-09; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Minimal Flow Anesthesia; Low Flow Anesthesia; Robotic Assisted Laparoscopic Abdominal Surgery
MeSH Terms: interventions — Blood Gas Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — blood gas analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: After intubation, a fresh gas flow of 3 L/min will be applied for the first 20 minutes and then reduced to 0.5 L/min.
  Interventions: Other: blood gas analysis
- Group 2: After intubation, a fresh gas flow of 3 L/min will be applied for the first 20 minutes and then reduced to 1 L/min.
  Interventions: Other: blood gas analysis

INTERVENTIONS:
Other: blood gas analysis — 1. Airway pressure (P plateau, Ppeak) values are taken from the anesthesia device data,
  2. BIS (from routine BIS monitoring)
  3. Temperature (routinely from pharyngeal temperature probe),
  4. Oxygen saturation (routinely from the patient monitor)
  5. End-tidal CO₂,
  6. inspiratory O₂ concentration,
  7. Inspiratory CO2 concentration,
  8. inspiratory and expiratory desflurane concentrations,
  9. tidal volume,
  10. MAC is routinely obtained from anesthesia device data.
  11. Blood Gas Analysis (COHgb, Ph, PO2, PCO2, SaO2, HCO3, Base deficit, glucose, lactate)

SUMMARY:
This study aims to compare the use of low fresh gas flow (1 L/min) desflurane anesthesia with minimum fresh gas flow (0.5 L/min) desflurane anesthesia in patients undergoing robotic-assisted abdominal surgery. The comparison will be based on hemodynamic and respiratory parameters. The secondary aim of our study is to compare the two different fresh gas flow methods in terms of inhalation agent consumption and soda lime consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robotic-assisted abdominal surgery

Exclusion Criteria:

* serious cardiac, respiratory, hepatic, renal, or mental disorders;
* hearing problems;
* anxiety, depression, or other psychiatric conditions;
* patient's request to leave the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing robotic-assisted abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
inspiratory O2 concentration | from beginning of anesthesia induction to the end of anesthesia (during periopertaive period)
  inspiratory O2 concentration is measured from anesthesia machine monitor
partial oxygen pressure | from beginning of anesthesia induction to the end of anesthesia (during periopertaive period)
  PO2 from blood gas analysis

SECONDARY OUTCOMES:
desflurane consumption | 3th hour
  desflurane consumption
changes in liver and kidney function tests from the preoperative values to 48 hours postoperative | postoperative 1st day
  to determine the changes in serum aspartate aminotransferase (AST), alanine aminotransferase (ALT), blood urea nitrogen (BUN), and creatinine from the preoperative values to 48 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Betül Güven Aytaç, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided